CLINICAL TRIAL: NCT06620341
Title: Comparing the Rate of Antibiotic Infusion Among Patients with Acute Upper Respiratory Tract Bacterial Infections in the Emergency Department -- a Cluster Randomized Controlled Trial
Brief Title: A Cluster Randomized Controlled Trial to Compare the Rate of Antibiotic Infusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-0469
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Acute Upper Respiratory Tract Infection; Bacterial Infections
Keywords: Bacterial infection of upper respiratory tract; Infusion rate; pharmacist
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Because of the nature of the intervention, masking of doctors and participants was not possible, but telephone follow-up staff and data analysts were masked to allocation group until after the definitive analysis was done.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacist medication education group (Experimental): Pharmacists give emergency doctors medication education every month about how to use antibiotic infusion reasonably
  Interventions: Behavioral: drug education
- No pharmacists' education on antibiotics (No Intervention): Following routine clinical practices, with no pharmacists' education on rational use of antibiotics

INTERVENTIONS:
Behavioral: drug education — * Training: Train emergency doctors every month on how to use antibiotic infusion reasonably; The prescription, cancellation, or method of use of antibiotics is decided by doctors.
    * Implementation of intervention cards: When the C-reactive protein (CRP) of patients is exceed 10mg/L, the doctor should determine whether to use antibiotics based on the clinical status of patients.
      * Promotion: Promote reasonably use of intravenous antibiotics through public accounts and posters.
        * Patient education: Distribute educational flyers to patients about how to use antibiotics reasonably.
  Arms: Pharmacist medication education group

SUMMARY:
Acute upper respiratory tract infection, commonly known as upper respiratory infection, is an acute inflammation primarily affecting the nose, pharynx, or larynx caused by various viruses and/or bacteria. Viruses are more common, accounting for 70% to 80% of cases, while bacterial infections account for 20% to 30%. For a long time, the high rate of intravenous infusion use has been a prominent issue in clinical diagnosis and treatment in China. The irrational and excessive use of antimicrobials in emergency patients with upper respiratory tract bacterial infections has also become increasingly apparent, imposing unnecessary financial burdens and risks of drug side effects on patients. Therefore, reducing the rate of intravenous antimicrobial administration in emergency patients with upper respiratory tract bacterial infections has become an urgent problem to be solved. By implementing measures such as health education by clinical pharmacists and enhancing the awareness of rational antimicrobial use in doctors, it is expected to lower the rate of intravenous antimicrobial administration, reduce the occurrence of drug resistance, improve treatment convenience for patients, and lower treatment costs while ensuring therapeutic efficacy.

The purpose of this study was to investigate whether clinical pharmacists can reduce the intravenous infusion rate of antimicrobials in emergency patients with upper respiratory tract bacterial infections through medication education for emergency medical staff and to observe whether this intervention will affect the prognosis and medication safety of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper respiratory tract infections seeking emergency medical attention;

  * Patients with laboratory tests indicating White Blood Cell (WBC) >10×10^9/L or White Blood Cell (CRP) ≥ 10.0mg/L, requiring the use of antimicrobial agents;

    * Patients aged ≥ 18 years; ④ Patients with at least one of the following local signs and symptoms: (1) fever, (2) cough, (3) rhinitis (sneezing, nasal congestion, or rhinorrhea), (4) pharyngitis (sore throat), (5) shortness of breath, (6) wheezing, (7) chest pain, (8) abnormal auscultation findings.

Exclusion Criteria:

* Patients with other infections in addition to upper respiratory tract infections; ② Patients who require hospitalization or treatment in a higher-level medical institution as assessed by medical professionals;

  * Patients who cannot take oral medications or have severe gastrointestinal dysfunction; ④ Special patients, including those with neutropenia, bone marrow suppression, during radiochemotherapy, undergoing immunosuppressive therapy, human immunodeficiency virus (HIV)-positive patients, patients with congenital immune deficiency, pregnant patients, and patients with mental illnesses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11900 (Estimated)
Dates: Start 2024-11-18 (Estimated); Primary Completion 2025-04-17 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Infusion rate of antibacterial drugs in patients with bacterial infection of upper respiratory tract | Through study completion, an average of 6 months

SECONDARY OUTCOMES:
Disease maintenance | Within 14 days after enrolment
  Days of respiratory tract infection symptoms keeps
Adverse drug reaction | Within 14 days after enrolment
  Allergic reaction, rash or pruritus
Disease recurrence within a 14 days period | Within 14 days after enrolment
  Patients re-attend outpatient clinic or emergency department of the hospital for treatment
Disease recurrence within a 14 days period | Within 14 days after enrolment
  Patients who did not re-attend outpatient clinic or emergency but re-used antibiotic infusion after first visit in emergency
Worsening of disease within a 14 days period | Within 14 days after enrolment
  Patients be hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Haibin Dai, Professor, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China